CLINICAL TRIAL: NCT00344565
Title: Combined Treatment of Modafinil and Cognitive Behavioral Therapy for Cocaine Dependence
Brief Title: A Placebo-Controlled Double-Blind Combined Treatment of Modafinil and CBT for Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Efrat Aharonovich, Research Scientist, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: # 5148; K23DA016743-03 (NIH)
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo, was matched to modafinil up to 400 mg/day. Patients also receive motivational interviewing and Cognitive Behavioral Therapy-Relapse Prevention (CBT-RP)
  Interventions: Drug: Modafinil; Behavioral: Cognitive Behavioral Therapy--Relapse Prevention
- Modafinil (Active Comparator): Modafinil (Active comparator). Patients received motivational interviewing and Cognitive Behavioral Therapy--relapse prevention (CBT-RP)
  Interventions: Drug: Modafinil; Behavioral: Cognitive Behavioral Therapy--Relapse Prevention

INTERVENTIONS:
Drug: Modafinil — During the first lead-in week, participants will attend the clinic 3 times per week, participate in one session of neuropsychological assessment and receive motivational interviewing and Cognitive Behavioral Therapy--Relapse Prevention (CBT-RP). At the end of the first lead-in week participants will be randomized to modafinil or placebo stratified by the levels of cocaine use, and whether or not abstinence was achieved. Participants will then be followed for 11 weeks with measures of cocaine cravings and withdrawal, and drug use outcome, and will receive CBT-RP.
  Other Names: Provigil
Behavioral: Cognitive Behavioral Therapy--Relapse Prevention — Once weekly individual session of motivational interviewing and Cognitive Behavioral Therapy--Relapse Prevention (CBT-RP)
  Other Names: CBT-RP

SUMMARY:
The purpose of this study is to test whether a cognitive behavioral therapy (CBT) and a medication called modafinil, which is approved to treat sleep disorders, will help individuals who are abusing cocaine.

DETAILED DESCRIPTION:
Chronic cocaine abuse has been documented to produce cognitive impairments in various domains. The observed cognitive deficits in the substance abuse population include, but are not restricted to, attention, concentration, verbal and nonverbal memory, problem solving and abstract reasoning. Our recent studies (IRB Protocol # 3998) demonstrated that in cocaine dependent participants such cognitive deficits have been shown to: 1) negatively effect retention and 2) impede the ability of the drug abuser to benefit from cognitive behavioral therapy- relapse prevention (CBT-RP) that requires participant to attend to novel stimuli, integrate new information with existing stores, and translate information into behavior change (Aharonovich, Hasin & Nunes, 2003; Aharonovich et al, in press). Furthermore, the toxic effects of cocaine together with withdrawal symptoms, such as fatigue and hypersomnia make it difficult to fully engage in any psychosocial intervention including CBT-RP.

Recent findings indicate that cocaine dysregulates reward-related glutamate pathways (Dackis & O'Brien, 2003; Kalivas et al, 2003). Modafinil is a medication known to improve attention, increase wakefulness, energy, and alertness in part by increasing glutamate levels. In light of this work and the negative affect of cognitive impairments on treatment outcomes, testing cognitive enhancing medications that act on glutamate pathways is a novel promising strategy for improving treatment for cocaine dependence. Modafinil is approved for sleep disorders and is a relatively safe medication for cocaine-dependent participants as it has a low abuse potential and has shown promise in a double blind placebo controlled trial for cocaine dependence (Rush et al, 2002; Jasinski, 2000, Dackis et al, 2005). We therefore propose a double blind placebo controlled 12-week exploratory pilot study of modafinil, a "wakefulness agent," in conjunction with sessions of CBT-RP enhanced with motivational interviewing components.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM IV criteria for current cocaine dependence and is seeking treatment.
* Used cocaine at least eight days in the past month or reports episodic binges of large amounts of cocaine (at least $150 worth) at least twice per month
* Able to give informed consent and comply with study procedures.

Exclusion Criteria:

* Meets DSM IV criteria for current mood disorder or past or current mania (i.e. bipolar disorder), schizophrenia or any psychotic disorder other than transient psychosis due to drug abuse.
* Baseline 21 item Hamilton Depression Scale scores ≥ 15
* History of seizures
* Chronic organic mental disorder.
* Significant current suicidal risk.
* Pregnancy, lactation, or failure in sexually active female participants to use adequate contraceptive methods.
* Unstable physical disorders, which might make participation hazardous such as hypertension, hepatitis, participants with mildly elevated AST and ALT levels (< 3 X upper limit or normal are acceptable), or diabetes.
* Coronary vascular disease as indicated by history, or suspected by abnormal EKG or history of cardiac symptoms.
* Current use of prescribed psychotropic medications.
* Current use of medications that interact with modafinil: Tricyclic anti-depressants; MOA Inhibitors; diazepam; phenytoin and medications containing Ethinyl Estradiol
* Known hypersensitivity to modafinil
* Currently meets DSM-IV criteria for narcolepsy
* Currently meets DSM-IV criteria for ADHD
* Currently meets DSM-IV criteria for opioid or sedative-hypnotic dependence.
* Currently meets criteria for DSM-IV alcohol dependence with evidence of clinically significant physiological dependence in need of medically supervised detoxification.
* Current cannabis dependence is identified as the main problem-i.e. participants with current DSM-IV cannabis dependence are eligible, as long as cocaine is identified by the participant as the primary substance problem for which they are seeking treatment.
* Gross visual or auditory impairments
* First language is not English and received NO formal education in English-speaking school

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Cocaine use outcome at week 12 (measured with urine toxicology and self-reports) | At week 12

SECONDARY OUTCOMES:
Cognitive functioning at week 12 (measured with neuropsychological assessment) | At week 12
Cocaine withdrawal symptoms throughout (measured with clinical assessments and self-reports) | At week 12

CONTACTS AND LOCATIONS:
Overall Officials: Efrat Aharonovich, PhD, Principal Investigator — Columbia University - New York State Psychiatric Institute